CLINICAL TRIAL: NCT04797767
Title: A Phase 1/2 Single-Center Trial Combining Venetoclax With G-CSF, Cladribine, Cytarabine, and Mitoxantrone (CLAG-M) for Patients With AML and High-Grade Myeloid Neoplasms
Brief Title: Venetoclax and CLAG-M for the Treatment of Acute Myeloid Leukemia and High-Grade Myeloid Neoplasms
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1121403; NCI-2021-01379 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10793 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Acute Biphenotypic Leukemia; Acute Myeloid Leukemia; Mixed Phenotype Acute Leukemia; Myeloid Neoplasm; Relapsed Acute Biphenotypic Leukemia; Relapsed Acute Myeloid Leukemia; Relapsed Mixed Phenotype Acute Leukemia; Relapsed Myeloid Neoplasm; Refractory Acute Biphenotypic Leukemia; Refractory Acute Myeloid Leukemia; Refractory Mixed Phenotype Acute Leukemia; Refractory Myeloid Neoplasm; Recurrent Myeloid Sarcoma
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute; Sarcoma, Myeloid | interventions — Cladribine; Cytarabine; Mitoxantrone; pegylated granulocyte colony-stimulating factor; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CLAG-M, venetoclax) (Experimental): Patients will receive induction with granulocyte colony-stimulating factor on days 0-5 (if peripheral white blood cell count is less than 20,000/uL), cladribine on days 1-5, cytarabine on 1-5, and mitoxantrone on days 1-3. Patients also receive venetoclax orally (PO) on days 1-14. Treatment repeats every 28-35 days for up to 2 induction cycles including mitoxantrone, and up to 4 consolidation cycles without mitoxantrone in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy and/or aspiration, and blood sample collection throughout the study.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Mitoxantrone; Biological: Recombinant Granulocyte Colony-Stimulating Factor; Drug: Venetoclax; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Mitoxantrone — Given IV
  Other Names: Dihydroxyanthracenedione; Mitozantrone
Biological: Recombinant Granulocyte Colony-Stimulating Factor — Given subcutaneously
  Other Names: Recombinant Colony-Stimulating Factor 3; rhG-CSF
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection

SUMMARY:
This phase I/II trial finds the best dose, side effects and how well giving venetoclax in combination with cladribine, cytarabine, granulocyte colony-stimulating factor, and mitoxantrone (CLAG-M) in treating patients with acute myeloid leukemia and high-grade myeloid neoplasms. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Chemotherapy drugs, such as cladribine, cytarabine, and mitoxantrone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving venetoclax with CLAG-M may kill more cancer cells.

DETAILED DESCRIPTION:
OUTLINE:

This is a dose-escalation study of venetoclax.

Patients will receive induction with granulocyte colony-stimulating factor subcutaneously (SC) on days 0-5 (if peripheral white blood cell count is less than 20,000/uL), cladribine intravenously (IV) on days 1-5, cytarabine IV on days 1-5, and mitoxantrone IV on days 1-3. Patients also receive venetoclax orally (PO) on days 1-14. Treatment repeats every 28-35 days for up to 2 induction cycles including mitoxantrone, and up to 4 consolidation cycles without mitoxantrone in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy and/or aspiration, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (per the World Health Organization [WHO] 2016 classification) or high-grade myeloid neoplasm (>= 10% myeloid blasts in peripheral blood or marrow as assessed by morphology or multiparameter flow cytometry at initial presentation). Patients with biphenotypic or mixed phenotype acute leukemia are eligible.
* PHASE I:

  * Newly diagnosed patients presenting for trial entry must have adverse risk disease as per the European LeukemiaNet 2017 guidelines
  * Relapsed/refractory patients presenting for trial entry must require first or subsequent salvage therapy and have detectable blasts in peripheral blood or >= 5% blasts in bone marrow, as assessed by morphology or multiparameter flow cytometry; or extramedullary myeloid sarcoma, per European LeukemiaNet 2017 guidelines.
  * These patients are only allowed in the phase 1 portion of the trial
* PHASE II: Newly diagnosed patients presenting for trial entry must have adverse risk disease as per the European LeukemiaNet 2022 guidelines
* Age >= 18 years
* Aspartate transaminase (AST) and alanine transaminase (ALT) =< 3.0 X upper limit of normal (ULN)
* Bilirubin =< 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
* Subject must have adequate renal function as demonstrated by a creatinine clearance >= 30 mL/min; calculated by the Cockcroft Gault formula or measured by 24 hours urine collection
* Left ventricular ejection fraction (LVEF) >= 45%, assessed by multigated acquisition (MUGA) or echocardiogram (ECHO) within 3 months prior to study day 0 or after most recent anthracycline administration if appropriate and no clinical evidence of congestive heart failure
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Treatment-related mortality (TRM) score < 13.1
* Female subjects of childbearing potential must have negative results for pregnancy test. Female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use an effective method of birth control from the time of signing the consent form until at least 3 months after the last dose of study drug
* Ability to understand and the willingness to sign a written informed consent document
* White blood cell count in peripheral blood must be < 25,000/ul prior to initiation of study therapy (CLAG-M plus venetoclax). Cytoreduction with hydroxyurea and/or cytarabine (e.g., 500 mg/m^2 per dose) is allowed to decrease the risk of tumor lysis syndrome

Exclusion Criteria:

* Acute promyelocytic leukemia or chronic myeloid leukemia in myeloid blast crisis
* Known active central nervous system (CNS) involvement with acute myeloid leukemia (AML)
* Concomitant illness associated with a likely survival of < 1 year
* Active systemic infection, unless disease is under treatment with antimicrobials and considered controlled or stable; patients with fever thought to be likely secondary to leukemia are eligible. Patients with chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment would be excluded. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface [HBs] antigen negative-, anti-HBs antibody positive and anti-hepatitis B core [HBc] antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate
* Known hypersensitivity to any study drug
* Pregnancy or lactation because of the unknown risks of this combination
* Concurrent treatment with any other investigational agent
* Subject is known to be positive for human immunodeficiency virus (HIV)
* Subjects who cannot discontinue concomitant CYP3A inhibitors, except for voriconazole, prior to cycle 1 day 1 (C1D1)
* Treatment with any of the following within 7 days prior to the first dose of venetoclax

  * Steroid therapy for anti-neoplastic intent
* Administration or consumption of any of the following within 3 days prior to the first dose of venetoclax:

  * Grapefruit or grapefruit products
  * Seville oranges (including marmalade containing Seville oranges)
  * Star fruit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (Phase I) | Up to 12 months
Maximum tolerated dose of venetoclax in combination with CLAG-M (Phase I) | Up to 12 months
Event free survival (Phase II) | At 6 months

SECONDARY OUTCOMES:
Complete remission rate | After 2 cycles (each cycle is approximately 35 days)
Rate of minimal residual disease negativity | Up to 1 year
Rate of allogeneic hematopoietic cell transplant | At 1 year
Overall survival | At 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Beth M. Percival, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raychaudhuri S, Gooley TA, Rasmussen A, Quach K, Gill E, Halpern AB, Appelbaum JS, Ghiuzeli CM, Hendrie PC, Cassaday RD, Walter RB, Percival MM. Phase 1 trial of venetoclax with cladribine, cytarabine, G-CSF, and mitoxantrone for AML and high-grade myeloid neoplasm. Blood Neoplasia. 2025 Mar 3;2(3):100085. doi: 10.1016/j.bneo.2025.100085. eCollection 2025 Aug. PMID 40535475